CLINICAL TRIAL: NCT01438684
Title: Phase 1 Study of RPh201 in Patients With Chronic Vegetative or Minimal Conscious State
Brief Title: The Impact of RPh201 on Chronic Vegetative State (CVS): fMRI Study
Acronym: RPh-in-CVS
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: due to lack of supply of medication and technical problems with the MRI
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 026011- HMO-CTIL
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2017-08

CONDITIONS: Chronic Vegetative State
Keywords: chronic vegetative state; functional MRI
MeSH Terms: conditions — Persistent Vegetative State | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- RPh201 group (Active Comparator): 7 patients will receive the treatment
  Interventions: Drug: RPh201
- non RPh201 group (Placebo Comparator): 3 patients will receive placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: RPh201 — 400 microliter s.c. twice a week for 3 months
  Arms: RPh201 group
Drug: Saline — 400 microliter Saline solution s.c. twice a week for 3 months
  Arms: non RPh201 group

SUMMARY:
The aim is to evaluate the impact of RPh201 on brain activity in chronic vegetative state patients. The assessment will be done using clinical measurements and functional MRI studies.

ELIGIBILITY:
Inclusion Criteria:

* chronic vegetative state patients

Exclusion Criteria:

* allergic reaction to treatment
* patients that can not undergo MRI
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-09; Primary Completion 2019-01 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
consciousness level measured clinically | 6 months
  Each patient will undergo a behavioral assessment (using the Coma Recovery Scale Revised) before treatment and every 2 weeks during the treatment period as well as 3 months following the end of the treatment. Complete blood counts, electrolytes, liver function tests, renal function tests and ECG will be performed every two weeks.

SECONDARY OUTCOMES:
Functional magnetic resonance imaging of cortical activity | 6 months
  3 scans will be performed: before treatment, after three months of treatment and 3 months after cessation of treatment. Scanning sessions will include a hierarchical auditory paradigm, an imagery task and resting state fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- Netta Levin, Jerusalem, Israel